CLINICAL TRIAL: NCT04038879
Title: Comparison Study of Echocardiography and Cardiovascular Magnetic Resonance Imaging in the Assessment of Mitral and Aortic Regurgitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Seth Uretsky, Medical Director, Cardiovascular Imaging, Atlantic Health System
Other Study IDs: 555087
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Mitral Regurgitation; Aortic Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mitral/Aortic Regurgitation: Subjects identified with mitral or aortic regurgitation will be asked to undergo testing with trans thoracic echocardiogram, stress echocardiography, and cardiac MRI with and without contrast. In addition, patients will be asked to answer the KCC and EQ5DL questionnaires.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI of the heart

SUMMARY:
The primary treatment for patients determined to have severe aortic or mitral regurgitation is surgical repair or replacement their valves. The most commonly used tool to quantify the severity mitral and aortic regurgitation is echocardiography. Studies have shown that echocardiography may have significant limitations in quantifying regurgitant volume. MRI has recently been shown to easily and reproducibly quantify regurgitation. To better understand how to accurately quantify severity of regurgitation the investigators propose this study with the following aims: 1) compare MRI to echocardiography in the evaluation of regurgitant volume in patients with aortic or mitral regurgitation and 2) to assess which technique is better at predicting the response of the left ventricle to valve surgery.

DETAILED DESCRIPTION:
The primary treatment for patients determined to have severe aortic or mitral regurgitation is surgical repair or replacement their valves. The most commonly used tool to quantify the severity mitral and aortic regurgitation is echocardiography. Studies have shown that echocardiography may have significant limitations in quantifying regurgitant volume. MRI has recently been shown to easily and reproducibly quantify regurgitation. To better understand how to accurately quantify severity of regurgitation the investigators propose this study with the following aims: 1) compare MRI to echocardiography in the evaluation of regurgitant volume in patients with aortic or mitral regurgitation and 2) to assess which technique is better at predicting the response of the left ventricle to valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Able to give informed consent
* Referred for isolated aortic or mitral valve repair or replacement due to valve regurgitation

Exclusion Criteria:

* Inability to provide consent.
* Pregnancy
* Claustrophobia
* Metallic contraindications to MRI (e.g. noncompatible aneurysm clip etc)
* Known intracardiac shunt
* Planned concomitant cardiac surgical procedure such as coronary artery bypass, septal myomectomy, or other valve procedure.
* More than mild mitral or aortic stenosis.
* For patients enrolled with mitral regurgitation: greater than mild aortic regurgitation.
* For patients enrolled with aortic regurgitation: greater than mild mitral regurgitation.
* Hypertrophic cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with mitral or aortic regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-07 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of echocardiography and MRI | 6 month
  Correlation of echocardiography and MRI
Change in LV EDV post surgery | 6 month
  Change in LV EDV post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uretsky S, Aldaia L, Marcoff L, Koulogiannis K, Hiramatsu S, Argulian E, Rosenthal M, Gillam LD, Wolff SD. The Effect of Systolic Variation of Mitral Regurgitation on Discordance Between Noninvasive Imaging Modalities. JACC Cardiovasc Imaging. 2019 Dec;12(12):2431-2442. doi: 10.1016/j.jcmg.2019.02.014. Epub 2019 Apr 17. PMID 31005539
- [Background] Uretsky S, Argulian E, Supariwala A, Marcoff L, Koulogiannis K, Aldaia L, Chaudhry FA, Wolff SD, Gillam LD. A Comparative Assessment of Echocardiographic Parameters for Determining Primary Mitral Regurgitation Severity Using Magnetic Resonance Imaging as a Reference Standard. J Am Soc Echocardiogr. 2018 Sep;31(9):992-999. doi: 10.1016/j.echo.2018.04.006. Epub 2018 Jun 18. PMID 29921479
- [Background] Uretsky S, Gillam L, Lang R, Chaudhry FA, Argulian E, Supariwala A, Gurram S, Jain K, Subero M, Jang JJ, Cohen R, Wolff SD. Discordance between echocardiography and MRI in the assessment of mitral regurgitation severity: a prospective multicenter trial. J Am Coll Cardiol. 2015 Mar 24;65(11):1078-88. doi: 10.1016/j.jacc.2014.12.047. PMID 25790878
- [Derived] Uretsky S, Gillam LD, Biederman RWW, Han Y, Jacob R, Martin ET, Langer M, Choi AD, Sultan I, Cavalcante JL, Shah DJ, Tong MS, Wolff SD, Sakul S, Guglielmo M, Pontone G. Sex differences in pre- and post-surgical left ventricular remodelling and outcomes in primary mitral regurgitation. Eur Heart J Cardiovasc Imaging. 2025 Jul 31;26(8):1429-1437. doi: 10.1093/ehjci/jeaf151. PMID 40392571
- [Derived] Uretsky S, Animashaun IB, Sakul S, Aldaia L, Marcoff L, Koulogiannis K, Argulian E, Rosenthal M, Wolff SD, Gillam LD. American Society of Echocardiography Algorithm for Degenerative Mitral Regurgitation: Comparison With CMR. JACC Cardiovasc Imaging. 2022 May;15(5):747-760. doi: 10.1016/j.jcmg.2021.10.006. Epub 2022 Jan 12. PMID 35324429
- [Derived] Uretsky S, Morales DCV, Aldaia L, Mediratta A, Koulogiannis K, Marcoff L, Sakul S, Wolff SD, Gillam LD. Characterization of Primary Mitral Regurgitation With Flail Leaflet and/or Wall-Impinging Flow. J Am Coll Cardiol. 2021 Dec 21;78(25):2537-2546. doi: 10.1016/j.jacc.2021.09.1382. PMID 34915984
- [Derived] Uretsky S, Aldaia L, Marcoff L, Koulogiannis K, Argulian E, Lasam G, Gillam L. Concordance and Discordance of Echocardiographic Parameters Recommended for Assessing the Severity of Mitral Regurgitation. Circ Cardiovasc Imaging. 2020 May;13(5):e010278. doi: 10.1161/CIRCIMAGING.119.010278. Epub 2020 May 15. PMID 32408828